CLINICAL TRIAL: NCT00984269
Title: Lymphedema Following Elective Hand and Wrist Surgery in Women Who Are Post Axillary Lymph Node Dissection: A Prospective, Randomized, Clinical Trial
Brief Title: Lymphedema Following Hand/Wrist Surgery in Women Post Axillary Node Dissection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-09-14B
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Tourniquet (No Intervention): Patients undergoing hand/wrist surgery without the use of a tourniquet.
- Tourniquet (Experimental): Patients undergoing hand/wrist surgery with the use of a tourniquet.
  Interventions: Procedure: Tourniquet Use

INTERVENTIONS:
Procedure: Tourniquet Use — Patients undergoing hand/wrist surgery with or without a tourniquet
  Arms: Tourniquet

SUMMARY:
This is a prospective, randomized, equivalence trial designed to evaluate postoperative complications following hand surgery with a brachial tourniquet and without a tourniquet in patients that have previously had a mastectomy with axillary node dissection with or without radiation treatment or history of lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of ipsilateral mastectomy with lymph node dissection with or without radiation treatment.
* Patients ages 18 and over
* Patients who have failed conservative, nonoperative treatment and present for an elective hand procedure with an anticipated tourniquet time of < 20 minutes.
* The subject is psychosocially, mentally, and physically able to understand and comply with the requirements of the study.

Exclusion Criteria:

* Patients that are not postoperative mastectomy with lymph node dissection with or without radiation treatment
* Patients under the age of 18
* Patients who are pregnant
* Patients presenting for an elective hand procedure with an anticipated tourniquet time of > 20 minutes.
* Patients who are on a blood thinner which cannot be stopped prior to surgery
* The subject has another concurrent physical or mental condition that is likely to affect compliance with the study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-08-19 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lymphedema 15% change from pre-post in girth | Preoperative,10-14 days, 6 weeks, 3 months, 6 months, and 1 year

SECONDARY OUTCOMES:
Wound assessment,Patient Satisfaction (on a scale of 0-10,Surgical and postoperative complications | 10-14 days, 6 weeks, 3 months, 6 months, and 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan Medical School, Ann Arbor, Michigan
  - OrthoCarolina, Charlotte, North Carolina